CLINICAL TRIAL: NCT06752928
Title: A Randomized Controlled Trial Comparing Dexcom Continuous Glucose Monitoring to Point of Care Glucose Testing for the Management of Hospital and Post-Discharge Subjects With Type 1 Diabetes
Brief Title: A Study Comparing Dexcom Continuous Glucose Monitoring to Point of Care Glucose Testing for the Management of Hospital and Post-Discharge Subjects With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008724
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: Continuous Glucose Monitoring; Type 1 Diabetes Mellitus; Point of Care
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Research design Adult subjects with T1D admitted to non-ICU medicine and surgery units and receiving insulin therapy will be randomized to either standard POC testing or Dexcom G7 CGM to guide insulin dose adjustments, with the POC group wearing a blinded CGM and the CGM group having insulin adjustments based on daily glucose profiles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Severe hyperglycemia will be managed by primary care professionals (Hospitalist Service) with intravenous or subcutaneous insulin therapy. Subjects will be invited to participate in the study after the resolution of severe hyperglycemia (BG < 400 mg/dl). Glucose monitoring by POC testing will be performed before meals and at bedtime. Results will be uploaded to the electronic medical record (EMR) system. The research team, together with the Primary care (PCP) team, will adjust daily insulin orders based on POC readings (standard of care). In addition, subjects will wear a 'blinded' CGM (no results will be visualized by patients, nursing staff, medicine, or research teams) during hospitalization for up to 10 days.
  Interventions: Diagnostic Test: Capillary Blood glucose Testing (POC)
- Dexcom CGM (Experimental): Severe hyperglycemia will be managed by primary care professionals (Hospitalist Service) intravenously with subcutaneous insulin therapy. Subjects will be invited to participate in the study after the resolution of severe hyperglycemia (BG < 400 mg/dl). Subjects will wear a real-time Dexcom G7 CGM for up to 10 days. Insulin therapy will be titrated based on daily CGM reports, including mean glucose, glycemic excursions, hypoglycemia, and severe hyperglycemia > 180 and >250 mg/dl values. Participants will wear a Dexcom rtCGM for up to 10 days during hospitalization.
  Interventions: Device: Dexcom G7 rtCGM

INTERVENTIONS:
Device: Dexcom G7 rtCGM — The Dexcom G7 Continuous Glucose Monitoring System (Dexcom G7 CGM System or G7) is a glucose monitoring system that continuously measures glucose in the interstitial fluid. It aids in the detection of episodes of hyperglycemia and hypoglycemia, facilitating both acute and long-term therapy adjustments
  Arms: Dexcom CGM
Diagnostic Test: Capillary Blood glucose Testing (POC) — POC glucose meters measure whole blood and convert the results to plasma glucose concentrations, which is the standardized form used in clinical practice.
  Other Names: POCT (point of care therapy)
  Arms: Standard of Care

SUMMARY:
This study aims to compare inpatient glycemic control by measuring the percentage of time in the range of 70-180 mg/dl and the frequency of hypoglycemia between Dexcom G7 Continuous Glucose Monitoring (CGM) and Point of Care (POC) Blood Glucose Testing in poorly controlled subjects with Type 1 Diabetes Mellitus.

The main question it aims to answer is:

-Whether there is a difference between POC testing (standard of care) and Real-time CGM in glycemic control and hypoglycemic events during hospitalization:

DETAILED DESCRIPTION:
The CDC reports that 1.6 million U.S. adults (5.7%) have type 1 diabetes (T1D), with hospitalization rates three times higher than the general population, primarily due to diabetes-related complications such as ketoacidosis and cardiovascular disease. A study at Emory University found that hospitalized T1D patients are younger, experience longer stays and more admissions, and face worse glycemic control and higher rates of hypoglycemia compared to type 2 diabetes (T2D) patients.

Point-of-care (POC) capillary glucose testing is the standard for monitoring hospitalized diabetes patients, but continuous glucose monitoring (CGM) offers more detailed glycemic profiles. Research, including trials using Dexcom CGM systems, has demonstrated CGM's superior ability to detect hypo- and hyperglycemia, reduce hypoglycemic events, and improve insulin therapy adjustments in T2D patients. However, no randomized controlled studies have evaluated the best glucose monitoring system for hospitalized T1D patients.

The proposed study aims to compare POC testing with Dexcom G7 CGM for guiding insulin therapy in hospitalized T1D patients. Researchers hypothesize that CGM will better prevent hypoglycemia and improve glycemic management during hospital stays, addressing a critical gap in evidence regarding glucose control's impact on T1D hospital outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Known history of T1D treated with insulin therapy (human regular or rapid-acting analogs or ultra-rapid analogs [lispro, aspart, glulisine, fast-acting insulin aspart, insulin lispro]), intermediate-acting (NPH and premixed formulations) or long-acting basal (glargine, detemir, degludec) formulations.
* Admission diagnosis of T1D with poorly controlled diabetes (blood glucose > 180 mg/dl, HbA1c > 7%), including diabetic ketoacidosis (DKA) and hyperglycemic hyperosmolar state (HHS).
* Expected length of hospital stay > three days at the time of randomization

Exclusion Criteria:

* Patients admitted to the ICU
* Subjects using CGM technology before admission
* Subjects with type 2 diabetes
* Treatment with systemic immunosuppressive agents
* Cystic fibrosis
* Prisoners
* Patients expected to require MRI procedures during hospitalization.
* Female subjects who are pregnant or breastfeeding at enrollment into the study.
* Subjects not willing to wear a CGM device
* Subjects with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension) and end-stage kidney disease (eGFR< 30 ml/min), or terminal illness.
* Subjects with a history of cognitive impairment, dementia, or mental condition rendering the subject unable to understand the nature and consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Through study completion (Day 10 or the length of admission)
  The total difference in blood sugar levels between the POC testing (standard of care) group and the rtCGM group throughout the hospitalization
Clinically significant hypoglycemia <54 mg/dl | Through study completion (Day 10 or the length of admission)
  The difference between blood sugar levels in POC testing (standard of care) group and rtCGM group during hospitalization

SECONDARY OUTCOMES:
Time above range | Through study completion (Day 10 or the length of admission)
  % time above Target Above range (TAR). Differences between the both groups will be calculated. (TAR, >250 mg/dl)
Time below range | Through study completion (Day 10 or the length of admission)
  % time in Below Target range (TBR). Differences between the both groups will be calculated.
  Differences between the both groups will be calculated. (TBR, < 70 and 54 mg/dl)
Glycemic Variability [% Coefficient of Variation (%CV) | Through study completion (Day 10 or the length of admission)
  % coefficient of variation will be measured during the intervention phase, compared to control, as measured by CGM.
Hypoglycemic events | Through study completion (Day 10 or the length of admission)
  Number of hypoglycemia events < 70 and 54 mg/dl
Hyperglycemic events | Through study completion (Day 10 or the length of admission)
  Number of hypoglycemia events >250 mg/dl
Nocturnal hypoglycemia | Through study completion (Day 10 or the length of admission)
  Number of hypoglycemic events (<70 and <54 mg/dl) between 22:00 and 06:00
Prolonged hypoglycemia | Through study completion (Day 10 or the length of admission)
  Number of events of Prolonged hypoglycemia < 70 mg/dl for more than 2 hours by CGM
Hospital Complications | Through study completion (Day 10 or the length of admission)
  Hospital complications include a composite of acute kidney injury (doubling of serum creatinine >0.5 mg/dl from baseline), cardiovascular events, infections, and death
Recurrent hypoglycemia | Through study completion (Day 10 or the length of admission)
  Number of recurrent hypoglycemic episodes (< 70 mg/dl)
Recurrent hyperglycemia | Through study completion (Day 10 or the length of admission)
  Number of recurrent hyperglycemic episodes (>250 mg/dl)

OTHER OUTCOMES:
Clinically significant hypoglycemia | Through study completion (Day 10 or the length of admission)
  Number of clinically significant hypoglycemic episodes: <54 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No